CLINICAL TRIAL: NCT01774500
Title: Study of Prognosis Value of Protein S100Beta and Copeptine in Seizure in the Emergency Department
Brief Title: Biomarkers In Seizure To Predict Recurrence and Severe Outcomes
Acronym: BISTRO
Status: Completed | Type: Observational
Sponsor: Bistro Study Group (Other)
Collaborators: Groupe Hospitalier Pitie-Salpetriere (Other); Barts & The London NHS Trust (Other)
Responsible Party: Principal Investigator, Yonathan Freund, Chef de Clinique - Research fellow. MD, Bistro Study Group
Other Study IDs: BISTRO
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Seizures; S-100b Protein; Copeptin
Keywords: biomarkers; Emergency Department; Seizures; epilepsy; S100b; copeptin
MeSH Terms: conditions — Seizures; Diabetes Insipidus; Emergencies; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — 2 5ml serum sample for proteine S100Beta and copeptine analysis

SUMMARY:
We study the hypothesis that combination of Proteine S100 beta and Copeptin within normal ranges can rule out seizure recurrences and severe outcome, and allow early discharge from the emergency department

DETAILED DESCRIPTION:
Prospective study for a 12 month period in Paris (France) and London (UK).

Inclusion criteria :

* seizure within 24h of attendance to an Emergency department (ED)
* or seizure in the ED

Exclusion Criterie :

* pregnancy
* prisoneer

Primary endpoint :

- recurrence of seizure, hospitalisation more than 24 hours or death within seven days

Secondary endpoint :

* Hospital free days at day 7 and day 28
* Death, ICU admission, or neurosurgical intervention at day 7 and day 28
* Return visit to the ED or re admission at day 7 and day 28

data collection:

* demographics
* past medical history, medication
* vital signs (Heart rate, temperature, Pulse oxymetry, blood pressure, GCS) on arrival
* Pathology (White cell count, Sodium, Calcium, Glucose, lactate)
* Protein S100B and Copeptin
* Seizure characteristics (Witnessed, simple, partial, complex, provoked, acute symptomatic, idiopathic)
* Discharge plan, outcomes

Follow up at day 7 and day 28, hospital visit or phone call

ELIGIBILITY:
Inclusion Criteria:

* Seizure within 24 hours of ED attendance
* Or Seizure in the ED

Exclusion Criteria:

* Pregnancy
* Prisoner
* age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency department patients
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Combined hospital admission, seizure recurrence, or death at day 7 | 7 days

SECONDARY OUTCOMES:
Hospital free days | 7 days
  number of days out of hospital, death corresponding to 0
Hospital free days | day 28
death or ICU admission | day 7
Death or ICU admission | 28 days
Recurrence of seizure | 7 days

CONTACTS AND LOCATIONS:
Locations (4):
- France (3):
  - Hopital Lariboisiere, Paris
  - Groupe Hospitalier pitie-salpetriere, Paris
  - Hopital Tenon, Paris
- Royal London Hospital, Barts Health NHS Trust, London, United Kingdom